CLINICAL TRIAL: NCT00203125
Title: Sub-study to Evaluate the Effect of An Oral Dose of Tyramine in Subjects Completing 26 Weeks of Participation in PRESTO (TVP-1012/133)
Brief Title: A Study to Evaluate the Effects of Tyramine in Patients Who Completed the PRESTO Study.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: J. Michael Nicholas, Sr. Director, US Regulatory Affairs, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVP - 1012/133a
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Tyramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rasagiline mesylate — 0.5 or 1 mg oral, once-daily
  Other Names: TVP-1012
Other: tyramine — 50 mg once daily

SUMMARY:
This study is to determine if Tyramine has any side effects on patients receiving 0.5mg, 1mg of Rasagiline or Placebo

ELIGIBILITY:
Inclusion Criteria:

Men and women with idiopathic Parkinson's disease (PD) who have met inclusion criteria for PRESTO, and have completed the 26-week PRESTO study. The subject should be available to participate in the sub-study immediately following the last PRESTO visit (same day). Subjects must continue PRESTO study drug until the morning of the Tyramine Sub-Study.

Subjects must provide separate informed consent to participate in the Tyramine Sub-Study.

Exclusion Criteria:

Subjects must not have a history of intracranial aneurysm or stroke.

Subjects should not have uncontrolled hypertension, defined as systolic pressure > 160 mmHg, or diastolic pressure > 90 mmHg.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2000-10; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
An increase in systolic blood pressure of > 30mmHg from the mean baseline value (documented by at least 3 consecutive measurements). Or Bradycardia with a heart rate below 40 beats per minute | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Salzman, Ph.D., Study Director — Teva Neuroscience, Inc.